CLINICAL TRIAL: NCT06130332
Title: A Single-center Exploratory Clinical Study of Neoadjuvant Tirellizumab Combined With Chemotherapy for Early Oral Squamous Cell Carcinoma (cT1-2N0M0)
Brief Title: Neoadjuvant Tirellizumab Combined With Chemotherapy for Early Oral Squamous Cell Carcinoma(HNC-SYSU-004)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-1064-01
Record Dates: First submitted 2023-11-01; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Oral Cancer; PD-1
MeSH Terms: conditions — Mouth Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 with chemotherapy (Experimental): Tirellizumab, Carboplatin,albumin-bound paclitaxel Patients receive Tirellizumab IV on day 1, albumin-bound paclitaxel IV on day 1 and carboplatin IV on day 1 . Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Then surgery.
  Intervention: Drug: Tirellizumab, Carboplatin, albumin-bound paclitaxel:2 cycles
  Surgery：Enlarged local excision，excision with the safe margin 1.0-1.5cm away from the original tumor
  Interventions: Drug: PD-1 with chemotherapy
- upright surgery (Other): Surgery：Primary resection，excision with the safe margin 1.0-1.5cm away from the original tumor
  selective neck dissection:I II III region neck dissection
  Interventions: Procedure: upright surgery

INTERVENTIONS:
Drug: PD-1 with chemotherapy — Tirellizumab+Carboplatin+albumin-bound paclitaxel:2 courses Tirellizumab,+Carboplatin+albumin-bound paclitaxel Tirellizumab (IV), dose= 200mg , day=1 , cycle length: 21 days. Carboplatin (IV), dose=300mg/m2, day= 1, cycle length: 21 days. albumin-bound paclitaxel (IV), dose=260mg/m2, day= 1, cycle length: 21 days.
  Intervention: Drug: Tirellizumab, Carboplatin, albumin-bound paclitaxel:2 cycles Surgery：Enlarged local excision，excision with the safe margin 1.0-1.5cm away from the original tumor
  Arms: PD-1 with chemotherapy
Procedure: upright surgery — Surgery：Primary resection，excision with the safe margin 1.0-1.5cm away from the original tumor
  selective neck dissection:I II III region neck dissection
  Arms: upright surgery

SUMMARY:
Surgery is usually the first choice for early-stage oral squamous cell carcinoma (OSCC). However, there is currently a lack of consensus on whether patients with clinically negative cervical lymph nodes (N0) should undergo elective neck dissection (END) at the same time. About 20-30% of cT1-2N0M0 oral cancer patients have occult lymph node metastasis, and existing examination methods cannot accurately predict occult cervical lymph node metastasis. Therefore, most clinical retrospective and prospective studies recommend END for cN0 patients. Previous studies have found that no cancer cells were found in the cervical lymph nodes of 70% of patients after END. This unselective END can cause patients with accessory nerve dysfunction, neck scars, etc., and prolong hospitalization and surgery time. Exploring the treatment model for patients with early-stage oral squamous cell carcinoma is an urgent problem that needs to be solved. This study intends to conduct a study on the neoadjuvant treatment of tislelizumab, carboplatin, and albumin-bound paclitaxel. After neoadjuvant immunotherapy in patients with early-stage oral cancer (T1-2N0M0), the primary tumor is treated with standard surgical treatment. Comparison with A single-center exploratory clinical study of traditional oral cancer radical resection + selective neck lymphadenectomy was conducted to explore its effectiveness through the difference in 2-year disease-free survival (DFS).

This research plan covers 40 patients with early-stage oral squamous cell carcinoma. They will be randomly divided into tislelizumab, chemotherapy combined with surgery (experimental group) and traditional surgery (control group) in a 1:1 ratio. The patients' tumors will be collected. Tissues, adjacent cancer tissues, whole blood samples, saliva samples, and matrix samples were used to observe the changes in imaging and pathology compared with treatment. At the same time, the clinical information of the patients was collected, such as quality of life indicators such as judgment function, pathological grading, staging, treatment, Spine, serology, imaging, etc., mainly to evaluate the 2-year event-free survival (EFS) between the experimental group and Weather Forecast, and the 3-year overall survival (OS) and patient quality of life between the experimental group and Weather Forecast.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early oral squamous cell carcinoma diagnosed as T1-2N0M0 according to the eighth edition of AJCC classification;
* No history of other malignant tumors;
* 18-75 years old;
* Baseline inspection is normal:

  1. The absolute value of neutrophil (ANC) ≥1.5x109/L in the past 14 days without the use of granulocyte colony-stimulating factor;
  2. Platelets ≥100×109/L without blood transfusion in the past 14 days;
  3. In the case of no blood transfusion or use of erythropoietin in the last 14 days, hemoglobin > 9g/dL;
  4. Total bilirubin ≤1.5× upper limit of normal (ULN);
  5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) in ≤2.5×ULN (patients with liver metastases allowed ALT or AST ≤5×ULN);
  6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min;
  7. Good coagulation function, defined as International standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
  8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
  9. The myocardial enzyme profile is within the normal range (if the researchers comprehensively judge that the simple laboratory abnormality is not clinically significant, it is also allowed to enter the group);
  10. For female subjects of reproductive age, a urine or serum pregnancy test should be performed within 3 days prior to receiving the first study drug administration (day 1 of cycle 1) and the result is negative. If the urine pregnancy test results cannot be confirmed as negative, a blood pregnancy test is requested. Women of non-reproductive age were defined as at least one year after menopause or having undergone surgical sterilization or hysterectomy;
  11. If there is a risk of conception, all subjects (male or female) are required to use contraception with an annual failure rate of less than 1% for the entire duration of treatment up to 120 days after the last study drug administration (or 180 days after the last chemotherapy drug administration).
* Sign informed consent.

Exclusion Criteria:

* Other malignant tumors are diagnosed, or oral cancer is not the beginning of neoadjuvant therapy;
* Prior to treatment, an active autoimmune disease requiring systemic treatment (such as the use of disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within the previous 2 years. Replacement therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
* known allogeneic organ transplantation (other than corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
* untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greater than the upper limit of normal value in the laboratory of the study center);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1. HBV viral load &lt before first dosing; 1000 copies /ml (200 IU/ml), subjects should receive anti-HBV therapy throughout study treatment to avoid viral reactivation;
2. For subjects with anti-HBC (+), HBsAg (-), anti-HBS (-) and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required;

   * active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
   * Pregnant or lactating women;
   * The presence of any serious or uncontrolled systemic disease, such as:

1) The resting electrocardiogram has major abnormal rhythm, conduction or morphology, such as complete left bundle branch block, heart block above Ⅱ degree, ventricular arrhythmia or atrial fibrillation; 2) Unstable angina pectoris, congestive heart failure, New York Heart Association (NYHA) grade ≥ 2 chronic heart failure;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  DFS(by months) is defined as the time from treatment until the date of the first relapse (local/regional recurrence or distant metastasis) or death (from any cause) whichever comes firsts and regardless of whether the patient withdraws from treatment or receives another anti-cancer therapy prior to disease DFS is defined as the time from treatment until the date of the first relapse (local/regional recurrence or distant metastasis) or death (from any cause) whichever comes firsts and regardless of whether the patient withdraws from treatment or receives another anti-cancer therapy prior to disease relapse.
Quality of life assessed by EORTC QLQ-H&N35. | 2 years
  The quality of life assessed by EORTC QLQ-H&N35(the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module-35)

SECONDARY OUTCOMES:
Overall survival(OS) | 5 years
  Overall survival(OS) is the time from day 1 of study treatment(the time randomized) until death from any cause.
Major pathologic response | 6 weeks
  Pathologic response rate to neoadjuvant treatment in resected tumor and lymph nodes. The rate of major pathologic response, defined as <10% residual viable tumor cells in the resection specimen will be compared to historic data with neoadjuvant chemotherapy.
Objective response rate, ORR | 6 weeks
  Objective tumor response, including CR and PR, was assessed using RECIST version 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen memorial hospital, Guangzhou, Guangdong, China